CLINICAL TRIAL: NCT06591559
Title: Up, Down, and All Around: Evaluating Mobility Devices for Young Children with Down Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Heather Feldner, Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00018915; 5TL1TR002318-07 (NIH)
Record Dates: First submitted 2024-06-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Down Syndrome
Keywords: early intervention; mobility aid; powered mobility; partial bodyweight support
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No Device (No Intervention): Children will play for 30 minutes using no mobility device.
- Explorer Mini in a Seated Posture (Active Comparator): Children will play for 30 minutes using the Explorer Mini a seated posture.
  Interventions: Device: Permobil Explorer Mini
- Explorer Mini in a Standing Posture (Active Comparator): Children will play for 30 minutes using the Explorer Mini a standing posture.
  Interventions: Device: Permobil Explorer Mini
- Portable Mobility Aid Partial Body Weight Support Harness (PUMA) (Active Comparator): Children will play for 30 minutes with partial bodyweight support provided by the PUMA.
  Interventions: Device: Portable Mobility Aid for Children (PUMA)

INTERVENTIONS:
Device: Permobil Explorer Mini — The Explorer Mini (Permobil AB, Sweden) is a commercially available, FDA approved powered mobility device intended for young children between 12-36 months of age with mobility limitations (weight limit: 35 lbs; height limit: 39.4 inches). It is lightweight (52 lbs. including battery) and fits in most automobiles (length: 25 inches; width: 19 inches; adjustable height: 29-37 inches). The Explorer Mini runs on a 12-volt battery with a driving range of 3.5 miles and a maximum speed of 1.5 mph, is controlled via a joystick with a 360-degree turning radius, has proportional speed control with 5 speed options, and can be used in a seated or standing position.
  Arms: Explorer Mini in a Seated Posture; Explorer Mini in a Standing Posture
Device: Portable Mobility Aid for Children (PUMA) — The Portable Mobility Aid for Children (PUMA; Enliten LLC) is a portable canopy system that utilizes an overhead support rail structure and a counterweight. The rail structure consists of two rigid parallel beams that mount to the canopy structure and one perpendicular mobile beam that allows for freedom of movement in one direction. Freedom of movement in the opposite direction is achieved by a system of pulleys along the movable beam that connects the harness to a counterweight. The counterweight provides a passive vertical force, counteracting gravity. The PUMA provides 2-dimensional mobility support over 81 ft2 (9 ft x 9 ft). The overhead bar is connected at 4 points to a child-worn harness. Children are free to move through many postures including sitting, crawling, standing, and walking.
  Arms: Portable Mobility Aid Partial Body Weight Support Harness (PUMA)

SUMMARY:
This research study will examine young children with Down syndrome's initial experiences with mobility devices. Children's biomechanics and exploration will be quantified while they are using both an overground partial bodyweight support system and powered mobility device.

DETAILED DESCRIPTION:
Young children with Down syndrome experience delays in cognition, communication, and mobility. As a result of cerebellar hypoplasia, children with Down syndrome have altered balance and coordination, muscle hypotonia, decreased muscle strength, and ligament laxity. Low muscle tone and ligament laxity can lead to the adoption of unfavorable postures, putting children at risk for developing musculoskeletal disorders in the future.

While children with Down syndrome are expected to walk, they do so significantly later than their peers, creating a gap in mobility, exploration, and socialization in the first years of life. Mobility during the first years is crucial to facilitate cascades of reciprocal development in cognition, communication, and motor skills, as well as reduce developmental delays and participation disparities for children with Down syndrome compared to their peers. While early intervention is common during this time to facilitate movement, clinical practice patterns vary widely and there are few evidence-based interventions or assistive technologies to support children and their families.

Treadmill training is currently the only intervention that has demonstrated efficacy for young children with hypotonia, but only for improving walking speed among already ambulatory children. Traditional treadmill training is limited, however, in that it does not allow for the sensorimotor experiences and social interactions that occur with self-initiated mobility in enriched, and often unpredictable, natural environments. As such, treadmill training and other clinical interventions may not fully address the need for holistic and multi-modal mobility opportunities.

Augmented mobility - in the form of partial bodyweight support systems, gait trainers, and powered mobility - has been proposed as a promising and complementary intervention to support early development in Down syndrome. While these tools have the potential to bridge the gap in self-initiated mobility and accelerate the onset of independent walking, little is scientifically known about how children engage with these devices nor how these devices shape their interactions with their environment. Furthermore, there is a lack of knowledge concerning the impact of different mobility devices on a child's physical development and posture.

In this research, the investigators propose to quantify a child's exploration, posture, and motor control strategies while using two promising assistive technologies for pre-ambulatory young children with Down syndrome: a partial-bodyweight support system (PUMA, Enliten, LLC.) and a powered mobility device (Explorer Mini, Permobil) that can be used in both seated and standing postures.

Participants will attend a total of four play sessions where they will play with a) no devices, b) partial bodyweight support, c) in the Explorer Mini in a standing posture, and d) in the Explorer Mini in a seated posture.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of Down syndrome
* are between 12-36 months of age
* are able to sit upright without support
* are able to tolerate moving through space while upright for 30 minutes
* are under 35 pounds in weight
* are under 39 inches tall in height

Exclusion Criteria:

* are able to walk 10 ft independently
* have had previous experience with the Explorer Mini or PUMA systems

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of space explored | At the end of each 30-minute play session for each study arm (session 1, session 2, session 3, session 4)
  The path of each child's movement during the play sessions will be tracked from video recordings and sensor data. The path will then be used to determine the percentage of the available play space that the child explored. Values will range from 0 - 100%, a higher value indicates more space explored.

SECONDARY OUTCOMES:
Normalized Integrated Electromyography (EMG) | At the end of each 30-minute play session for each study arm (session 1, session 2, session 3, session 4)
  Children will wear electromyography (EMG) sensors while playing. We will measure the bilateral muscle activity of the tibialis anterior, gastrocnemius, quadriceps, hamstrings (biceps femoris), erector spinae, and cervical paraspinal using surface EMGs. EMG data will be high-pass filtered (40 Hz), rectified, and low-pass filtered (10 Hz) to create a linear envelope of muscle activity during play sessions. For each muscle group, we will calculate the integrated EMG signal, or area under the curve, for each session normalized by time in device. Values will range from 0 to 100%, higher values indicate more muscle activity.
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) 2.1: Children Version | At the end of each 30-minute play session for each study arm (session 1, session 2, session 3, session 4)
  The QUEST 2.1: Children Version is an extension of the original QUEST tool tailored specifically for children who use assistive technology. The primary aim of this test is to evaluate how well assistive technology devices meet the needs of children and enhance their overall satisfaction with these devices. The questionnaire is designed to gather information on various aspects of the assistive technology, including its functionality, ease of use, and impact on the life of the user.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Feldner, PhD, PT, PCS, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No